CLINICAL TRIAL: NCT00706355
Title: Phase 1 Safety, Pharmacokinetic and Pharmacodynamic Study of PF-4217903 in Patients With Advanced Cancer
Brief Title: A Study of PF-04217903 in Patients With Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B0331002
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Results first posted 2012-05-31 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — 2-(4-(3-quinolin-6-ylmethyl-3H-(1,2,3)triazolo(4,5-b)pyrazin-5-yl)pyrazol-1-yl)ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: PF-04217903

INTERVENTIONS:
Drug: PF-04217903 — Escalating doses of PF-04217903 will be administered orally on a continuous dosing schedule. Doses to be evaluated will range from 50 mg BID to 1000 mg BID. A cycle is considered to be 21 days

SUMMARY:
PF-04217903 may work in cancer by blocking the cell growth, migration and invasion of tumor cells. PF-04217903 is a new member in a class of drugs called c-Met/hepatocyte growth factor receptor tyrosine kinase inhibitors. This research study is the first time PF-04217903 will be given to patients. PF-04217903 is taken by mouth daily.

DETAILED DESCRIPTION:
The study was prematurely discontinued due to a strategic development decision by Pfizer on 10FEB2012. The decision to terminate was not based on any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid tumors, histologically proven at diagnosis which is refractory to standard of care or for whom no standard of care therapy is available
* Adequate blood cell counts, normal kidney function, and performance status of 0 or 1

Exclusion Criteria:

* Major surgery, radiation therapy or anti-cancer therapy within 2 weeks of starting study treatment
* Prior stem cell transplant
* Active or unstable cardiac disease or heart attack within 12 months of starting study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Detroit, Michigan

REFERENCES:
- [Derived] Diamond JR, Salgia R, Varella-Garcia M, Kanteti R, LoRusso PM, Clark JW, Xu LG, Wilner K, Eckhardt SG, Ching KA, Lira ME, Schoenmakers EF, Christensen JG, Camidge DR. Initial clinical sensitivity and acquired resistance to MET inhibition in MET-mutated papillary renal cell carcinoma. J Clin Oncol. 2013 Jun 1;31(16):e254-8. doi: 10.1200/JCO.2012.46.4289. Epub 2013 Apr 22. No abstract available. PMID 23610116
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0331002&StudyName=A%20Study%20of%20PF-04217903%20in%20Patients%20with%20Advanced%20Cancer

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-04217903 50 mg: Two tablets 25 milligram (mg) PF-04217903 administered orally twice a day in continuous 21-day cycles.
- PF-04217903 100 mg: Four tablets 25 mg PF-04217903 administered orally twice a day in continuous 21-day cycles.
- PF-04217903 200 mg: One tablet 125 mg and 3 tablets 25 mg PF-04217903 administered orally twice a day in continuous 21-day cycles.
- PF-04217903 150 mg: One tablet 125 mg and 1 tablet 25 mg PF-04217903 administered orally twice a day in continuous 21-day cycles.
Period: Period 1: PF-04217903 50 mg
Arm/Group | PF-04217903 50 mg | PF-04217903 100 mg | PF-04217903 200 mg | PF-04217903 150 mg
Started | 3 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Objective progression or relapse | 2 | 0 | 0 | 0
Period: Period 2: PF-04217903 100 mg
Arm/Group | PF-04217903 50 mg | PF-04217903 100 mg | PF-04217903 200 mg | PF-04217903 150 mg
Started | 0 | 7 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 7 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Global deterioration of health status | 0 | 1 | 0 | 0
Not completed — Objective progression or relapse | 0 | 5 | 0 | 0
Period: Period 3: PF-04217903 200 mg
Arm/Group | PF-04217903 50 mg | PF-04217903 100 mg | PF-04217903 200 mg | PF-04217903 150 mg
Started | 0 | 0 | 2 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Period: Period 4: PF-04217903 150 mg
Arm/Group | PF-04217903 50 mg | PF-04217903 100 mg | PF-04217903 200 mg | PF-04217903 150 mg
Started | 0 | 0 | 0 | 4
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 2
Not completed — Objective progression or relapse | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- PF-04217903 50 mg: Two tablets 25 mg PF-04217903 administered orally twice a day in continuous 21-day cycles.
- Total: Total of all reporting groups
Arm/Group | PF-04217903 50 mg | PF-04217903 100 mg | PF-04217903 200 mg | PF-04217903 150 mg | Total
Number analyzed (Participants) | 3 | 7 | 2 | 4 | 16
Age Continuous [Mean (Standard Deviation); unit: Years] | 71.3 (8.6) | 50.6 (10.8) | 66.0 (18.4) | 54.0 (13.9) | 57.3 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 1 | 6
  Male | 1 | 5 | 1 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: MTD: dose level at which 1 of 6 participants experienced dose-limiting toxicity (DLT) after 21 days of treatment (Cycle 1). DLT: grade (Gr) 2 elevated creatinine, acute renal failure, Gr 3 thrombocytopenia with bleeding, hypertension (if unmanageable),Gr >=3 non-hematological non-disease-related (NDR) toxicities (except alopecia,Gr 3/4 hypophosphatemia, hyperuricemia), Gr 3/4 nausea, vomiting, diarrhea, Gr 4 neutropenia, thrombocytopenia lasting for >=7 days, febrile neutropenia, neutropenic infection, inability to deliver 80 percent of planned dose during Cycle 1 due to NDR toxicities.
Time Frame: Baseline up to 21 days after the start of each increased treatment dose
Population: Analysis population included all enrolled participants who received at least 1 dose of the study treatment.
Measure: Number; unit: mg
Groups:
- All Treated Participants: All participants who received PF-04217903 tablet (50 mg, 100 mg, 200 mg and 150 mg) orally twice a day in continuous 21-day cycles.
Arm/Group | All Treated Participants
Number analyzed (Participants) | 16
mg | 100

2. Primary Outcome: Recommended Phase 2 Dose (RP2D)
Time Frame: Baseline up to 21 days after the start of each increased treatment dose
Population: Data was not analyzed due to insufficient number of participants enrolled.
Measure: Number; unit: mg
Arm/Group | All Treated Participants
Number analyzed (Participants) | 0

3. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: DLT includes Gr 2 elevated creatinine and acute renal failure, Gr 3 thrombocytopenia with bleeding, hypertension (if unmanageable), Gr >= 3 non-hematological non-disease-related (NDR) toxicities (except alopecia, Gr 3/4 hypophosphatemia, hyperuricemia), Gr 3/4 nausea, vomiting, diarrhea, Gr 4 neutropenia, thrombocytopenia lasting for >= 7 days, febrile neutropenia, neutropenic infection, inability to deliver at least 80 percent of planned dose during Cycle 1 due to NDR adverse events.
Time Frame: Baseline up to 21 days after the start of each increased treatment dose
Population: DLT analysis set: participants who received first cycle of study medication and did not temporarily or permanently discontinue from study medication or missed more than 3 consecutive days of PF-04217903 dosing for reasons other than DLTs within first cycle.
Measure: Number; unit: Participants
Arm/Group | PF-04217903 50 mg | PF-04217903 100 mg | PF-04217903 200 mg | PF-04217903 150 mg
Number analyzed (Participants) | 3 | 7 | 2 | 4
Participants | 0 | 0 | 2 | 2

4. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for PF-04217903 and PF-04217903 Metabolite (PF-04328029)
Time Frame: 0 (pre-dose), 1, 2, 4, 6, 8 and 12 hours (hrs) (just prior to evening dosing) post dose on Cycle (C) 1 Day (D) 1 and C2 D1
Population: The pharmacokinetic (PK) parameter analysis population included all enrolled participants who received the study medication and had at least 1 of the PK parameters of interest. 'n' signifies those participants evaluated for this measure at specific time point for each arm group respectively.
Measure: Geometric Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | PF-04217903 50 mg | PF-04217903 100 mg | PF-04217903 200 mg | PF-04217903 150 mg
Number analyzed (Participants) | 3 | 7 | 2 | 4
Nanogram per milliliter (ng/mL)
  PF-04217903 (C1 D1) (n=3, 7, 2, 4) | 532.8 (90.598) | 397.0 (811.78) | 846.7 (1210.6) | 429.9 (942.74)
  PF-04217903 (C2 D1) (n=2, 4, 0, 2) | 663.4 (53.033) | 604.2 (347.62) | NA (NA) — Data was not analyzed as the participants did not receive the study treatment in this cycle. | 225.1 (66.468)
  PF-04328029 (C1 D1) (n=3, 7, 2, 4) | 105.6 (23.493) | 83.70 (95.953) | 203.0 (217.08) | 81.72 (132.71)
  PF-04328029 (C2 D1) (n=2, 4, 0, 2) | 113.9 (58.973) | 154.5 (89.706) | NA (NA) — Data was not analyzed as the participants did not receive the study treatment in this cycle. | 40.39 (14.354)

5. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin) for PF-04217903 and PF-04217903 Metabolite (PF-04328029)
Description: Participants did not receive 200 mg twice a day dose of study treatment for this specific measure.
Time Frame: 0 (pre-dose), 1, 2, 4, 6, 8 and 12 hrs (just prior to evening dosing) post dose on C2 D1
Population: The PK parameter analysis population included all enrolled participants who received the study medication and had at least 1 of the PK parameters of interest. 'n' signifies those participants evaluated for this measure at specific time point for each arm group respectively.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04217903 50 mg | PF-04217903 100 mg | PF-04217903 150 mg
Number analyzed (Participants) | 3 | 7 | 4
ng/mL
  PF-04217903 (n=2, 4, 2) | 0.0779 (42.851) | 34.72 (26.738) | 93.47 (86.621)
  PF-04328029 (n=2, 4, 2) | 0.0374 (9.8995) | 11.43 (8.7993) | 16.23 (15.825)

6. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) for PF-04217903 and PF-04217903 Metabolite (PF-04328029)
Time Frame: 0 (pre-dose), 1, 2, 4, 6, 8 and 12 hrs (just prior to evening dosing) post dose on C1 D1 and C2 D1
Population: as for outcome 5
Measure: Median (Full Range); unit: hr
Arm/Group | PF-04217903 50 mg | PF-04217903 100 mg | PF-04217903 200 mg | PF-04217903 150 mg
Number analyzed (Participants) | 3 | 7 | 2 | 4
hr
  PF-04217903 (C1 D1) (n=3, 7, 2, 4) | 1.00 [1.00 to 4.00] | 1.00 [1.00 to 4.33] | 1.03 [1.00 to 1.05] | 1.50 [1.00 to 4.00]
  PF-04217903 (C2 D1) (n=2, 4, 0, 2) | 1.00 [1.00 to 1.00] | 2.42 [1.00 to 4.00] | NA [NA to NA] — Data was not analyzed as the participants did not receive the study treatment in this cycle. | 2.50 [1.00 to 4.00]
  PF-04328029 (C1 D1) (n=3, 7, 2, 4) | 1.00 [1.00 to 4.00] | 1.00 [1.00 to 6.00] | 2.00 [2.00 to 2.00] | 1.50 [1.00 to 8.00]
  PF-04328029 (C2 D1) (n=2, 4, 0, 2) | 1.00 [1.00 to 1.00] | 2.42 [1.00 to 4.00] | NA [NA to NA] — Data was not analyzed as the participants did not receive the study treatment in this cycle. | 2.00 [0.00 to 4.00]

7. Secondary Outcome: Pre-dose Plasma Concentration (Ctrough) for PF-04217903 and PF-04217903 Metabolite (PF-04328029)
Description: Participants did not receive 200 mg twice a day dose of study treatment for this specific measure.
Time Frame: 0 (pre-dose), 1, 2, 4, 6, 8 and 12 hrs (just prior to evening dosing) post dose on C1 D1 and C2 D1
Population: The PK parameter analysis population included all enrolled participants who received the study medication and had at least 1 of the PK parameters of interest. 'n' signifies those participants evaluable for this measure.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04217903 50 mg | PF-04217903 100 mg | PF-04217903 150 mg
Number analyzed (Participants) | 3 | 7 | 4
ng/mL
  PF-04217903 (C1 D1) (n=3, 7, 4) | 0.0001 (0.0) | 0.0001 (0.0) | 0.0001 (0.0)
  PF-04217903 (C2 D1) (n=3, 6, 3) | 15.10 (29.413) | 3.705 (35.875) | 1.229 (92.147)
  PF-04328029 (C1 D1) (n=3, 7, 4) | 0.0001 (0.0) | 0.0001 (0.0) | 0.0006 (0.0670)
  PF-04328029 (C2 D1) (n=3, 6, 3) | 4.939 (7.4862) | 1.540 (10.524) | 0.4501 (26.340)

8. Secondary Outcome: Area Under the Plasma Concentration Time-curve From Zero to the Last Measured Concentration [AUC(0-last)] for PF-04217903 and PF-04217903 Metabolite (PF-04328029)
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast).
Time Frame: 0 (pre-dose), 1, 2, 4, 6, 8 and 12 hrs (just prior to evening dosing) post dose on C1 D1 and C2 D1
Population: as for outcome 5
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PF-04217903 50 mg | PF-04217903 100 mg | PF-04217903 200 mg | PF-04217903 150 mg
Number analyzed (Participants) | 3 | 7 | 2 | 4
ng*hr/mL
  PF-04217903 (C1 D1) (n=3, 7, 2, 4) | 1694.0 (254.23) | 1595.0 (1933.5) | 3005.0 (3125.4) | 1912 (2421.7)
  PF-04217903 (C2 D1) (n=2, 4, 0, 2) | 2003.0 (304.06) | 2308.0 (726.42) | NA (NA) — Data was not analyzed as the participants did not receive the study treatment in this cycle. | 1242 (505.58)
  PF-04328029 (C1 D1) (n=3, 7, 2, 4) | 384.7 (166.52) | 356.4 (249.31) | 1007.0 (1280.6) | 362.7 (426.32)
  PF-04328029 (C2 D1) (n=2, 4, 0, 2) | 404.2 (113.14) | 648.8 (261.85) | NA (NA) — Data was not analyzed as the participants did not receive the study treatment in this cycle. | 218.8 (100.41)

9. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval [AUC(0-tau)] for PF-04217903 and PF-04217903 Metabolite (PF-04328029)
Description: Area under the concentration-time profile from time zero to time tau (dosing interval), where tau is equal to 12 hours.
Time Frame: 0 (pre-dose), 1, 2, 4, 6, 8 and 12 hrs (just prior to evening dosing) post dose on C1 D1 and C2 D1
Population: as for outcome 5
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PF-04217903 50 mg | PF-04217903 100 mg | PF-04217903 200 mg | PF-04217903 150 mg
Number analyzed (Participants) | 3 | 7 | 2 | 4
ng*hr/mL
  PF-04217903 (C1 D1) (n=3, 7, 2, 4) | 1839.0 (311.34) | 1685.0 (2086.8) | 3320.0 (3217.3) | 2062 (2352.1)
  PF-04217903 (C2 D1) (n=2, 4, 0, 1) | 2178.0 (388.91) | 2516.0 (828.45) | NA (NA) — Data was not analyzed as the participants did not receive the study treatment in this cycle. | 1050 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  PF-04328029 (C1 D1) (n=3, 7, 2, 4) | 423.5 (197.62) | 378.7 (261.78) | 1214.0 (1599.5) | 390.0 (413.27)
  PF-04328029 (C2 D1) (n=2, 4, 0, 1) | 454.9 (101.12) | 722.3 (305.86) | NA (NA) — Data was not analyzed as the participants did not receive the study treatment in this cycle. | 179.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.

10. Secondary Outcome: Accumulation Ratio (Rac) for PF-04217903 and PF-04217903 Metabolite (PF-04328029)
Description: Rac is obtained from AUCtau (Cycle 2 Day 1) divided by AUCtau (Cycle 1 Day 1). Participants did not receive 200 mg twice a day dose of study treatment for this specific measure.
Time Frame: 0 (pre-dose), 1, 2, 4, 6, 8 and 12 hrs (just prior to evening dosing) post dose on C2 D1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | PF-04217903 50 mg | PF-04217903 100 mg | PF-04217903 150 mg
Number analyzed (Participants) | 3 | 7 | 4
Ratio
  PF-04217903 (n=2, 4, 1) | 1.097 (0.2871) | 2.413 (2.0866) | 1.040 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  PF-04328029 (n=2, 4, 1) | 0.9875 (0.2864) | 2.551 (2.4588) | 0.8660 (NA) — Standard deviation was not estimable since only one participant was evaluable.

11. Secondary Outcome: Metabolite to Parent Ratio Area Under the Curve From Time Zero to End of Dosing Interval (MRAUCtau)
Description: Molar ratio of metabolite to parent area under the plasma concentration time-curve from zero (pre-dose) to end of dosing interval (MRAUCtau).
Time Frame: 0 (pre-dose), 1, 2, 4, 6, 8 and 12 hrs (just prior to evening dosing) post dose on C1 D1 and C2 D1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | PF-04217903 50 mg | PF-04217903 100 mg | PF-04217903 200 mg | PF-04217903 150 mg
Number analyzed (Participants) | 3 | 7 | 2 | 4
Ratio
  C1 D1 (n=3, 7, 2, 4) | 0.2283 (0.0693) | 0.2297 (0.0759) | 0.3585 (0.0969) | 0.1828 (0.0148)
  C2 D1 (n=2, 4, 0, 1) | 0.2090 (0.0806) | 0.2790 (0.0413) | NA (NA) — Data was not analyzed as the participants did not receive the study treatment in this cycle. | 0.1650 (NA) — Standard deviation was not estimable since only one participant was evaluable.

12. Secondary Outcome: Apparent Oral Clearance (CL/F) for PF-04217903
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood. Participants did not receive 200 mg twice a day dose of study treatment for this specific measure.
Time Frame: 0 (pre-dose), 1, 2, 4, 6, 8 and 12 hrs (just prior to evening dosing) post dose on C2 D1
Population: The PK parameter analysis population included all enrolled participants who received the study medication and had at least 1 of the PK parameters of interest. 'N' (number of participants analyzed) signifies those participants evaluable for this measure.
Measure: Geometric Mean (Standard Deviation); unit: Liter/hr (L/hr)
Arm/Group | PF-04217903 50 mg | PF-04217903 100 mg | PF-04217903 150 mg
Number analyzed (Participants) | 2 | 4 | 1
Liter/hr (L/hr) | 22.97 (4.0305) | 39.71 (18.634) | 143.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.

13. Secondary Outcome: Change From Baseline in Tumor Proliferation Using F-Fluoro-3'-Deoxy-3'-L-Fluorothymidine Positron Emission Tomography (FLT-PET) Imaging at Day 1 of Cycle 2
Description: F-fluoro-3'-deoxy-3'-L-fluorothymidine positron emission tomography (FLT-PET) imaging was used to assess the tumor proliferation in RP2D cohorts. Results of the FLT-PET were scored according to the methods developed by the American College of Radiology Imaging Network (ACRIN).
Time Frame: Cycle 2 Day 1
Population: Data was not analyzed due to insufficient number of participants enrolled.
Measure: Mean (Standard Deviation); unit: Standardized Uptake Value (SUV)
Arm/Group | PF-04217903 50 mg | PF-04217903 100 mg | PF-04217903 200 mg | PF-04217903 150 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Secondary Outcome: Percentage of Participants With Objective Response (OR)
Description: Percentage of participants with OR based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed response were those that persisted on repeat imaging study at least 4 weeks after initial documentation of response. CR was defined as disappearance of all lesions (target and/or non target). PR were those with at least 30 percent decrease in sum of the longest dimensions of target lesions taking as a reference the baseline sum longest dimensions, with non target lesions not increased or absent.
Time Frame: Baseline until disease progression up to C2 D1
Population: Efficacy analysis set included all enrolled participants who received the study treatment and had measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PF-04217903 50 mg | PF-04217903 100 mg | PF-04217903 200 mg | PF-04217903 150 mg
Number analyzed (Participants) | 3 | 7 | 2 | 4
Percentage of participants | 0 [0.0 to 70.8] | 0 [0.0 to 41.0] | 0 [0.0 to 84.2] | 0 [0.0 to 60.2]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-04217903 50 mg | PF-04217903 100 mg | PF-04217903 200 mg | PF-04217903 150 mg
Serious Adverse Events (participants affected / at risk) | 0/3 | 3/7 | 1/2 | 2/4
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 2/2 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04217903 50 mg (N=3) | PF-04217903 100 mg (N=7) | PF-04217903 200 mg (N=2) | PF-04217903 150 mg (N=4)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04217903 50 mg (N=3) | PF-04217903 100 mg (N=7) | PF-04217903 200 mg (N=2) | PF-04217903 150 mg (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0
Atrophy (General disorders) | 0 | 0 | 0 | 1
Catheter site related reaction (General disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 1 | 1
Local swelling (General disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 2 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0
Performance status decreased (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 2 | 1 | 1
Blood glucose increased (Investigations) | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 1 | 0 | 0
Electrocardiogram ST segment depression (Investigations) | 1 | 0 | 0 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 1 | 0
Glucose urine present (Investigations) | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 2 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Insufficient number of participants had been enrolled in the study due to a strategic development decision; therefore some of the objectives for this study were either not investigated or not fully investigated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.